CLINICAL TRIAL: NCT04263792
Title: [18F]Fluoropropyl-Trimethoprim ([18F]F-TMP) PET/CT Imaging to Evaluate Biodistribution and Kinetics in Human Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833998
Record Dates: First submitted 2020-01-16; First posted 2020-02-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biodistribution cohort (Other): The Biodistribution cohort will include up to 5 patients who will undergo a series of vertex to mid-thigh (or feet if indicated) biodistribution [18F]fluoropropyl-trimethoprim PET/CT scans over a period of approximately 4 hours.
  Interventions: Drug: [18F]fluoropropyl-trimethoprim
- The Dynamic cohort (Other): The Dynamic cohort will include up to 15 patients who will undergo approximately 60 minutes of dynamic scanning followed by up to 2 static skull base to mid-thigh (or feet if indicated) scans post injection of [18F]fluoropropyl-trimethoprim.
  Interventions: Drug: [18F]fluoropropyl-trimethoprim

INTERVENTIONS:
Drug: [18F]fluoropropyl-trimethoprim — [18F]Fluoropropyl-Trimethoprim, also known as [18F]F-TMP, is a radiolabeled imaging agent for positron emission tomography (PET/CT).The use most relevant to this protocol is for imaging bacterial infection in human subjects. The parent compound, trimethoprim (TMP) is a well-known, safe, broad-spectrum, synthetic, small molecule antibiotic that has been used clinically for over 50 years for the treatment of acute bacterial infection and has been combined with sulfa-based antibiotics (Bactrim/Septra) for bacterial infection prophylaxis especially in the lung and bladder. An immediate clinical use for TMP radiotracers is imaging of pathologic bacteria that are the cause of human infection.

SUMMARY:
The purpose of this study is to study a radioactive tracer, a type of imaging drug that is injected into the body to see how it is taken up in sites of active infection using an imaging procedure called Positron Emission Tomography/Computed Tomography (PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Known or suspected bacterial infection, per clinical documentation of suspected infection (e.g. lab results, pathology results, physician progress notes, clinical symptoms of infection)
* Able to understand the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures

Exclusion Criteria:

* Antibiotic therapy with trimethoprim within 48h of the baseline PET/CT scan
* Inability to tolerate imaging procedures, in the opinion of an investigator or treating physician
* Unstable or other severe medical or psychological comorbidities that would compromise the subject's safety or successful participation in the study, in the opinion of an investigator or treating physician
* Pregnant or breast feeding patients; a urine pregnancy test will be performed in women of child-bearing potential prior to [18F]F-TMP injection, to confirm non-pregnant status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Understand the biodistribution of F-TMP in human patients by looking at the F-TMP uptake in PET/CT scans | 3 year
  Understand the biodistribution of F-TMP in human patients by comparing the F-TMP uptake using maxSUV and meanSUV of each ROI which will be drawn manually in tissues of interest including but not limited to: Blood pool, heart muscle, brain, thyroid, lymph nodes, lung, liver, kidney, small bowel, large bowel, adrenal gland, pancreas, gall bladder, bone, muscle, and gonads.
Understanding the kinetics of uptake of [18F]F-TMP in human patients by looking at the F-TMP uptake in PET/CT scans | 3 years
  Understanding the the kinetics of uptake of [18F]F-TMP in human patients by comparing the F-TMP uptake using maxSUV and meanSUV of each ROI which will be drawn manually in tissues of interest including but not limited to: Blood pool, heart muscle, brain, thyroid, lymph nodes, lung, liver, kidney, small bowel, large bowel, adrenal gland, pancreas, gall bladder, bone, muscle, and gonads.

SECONDARY OUTCOMES:
Compare the uptake of [18F]F-TMP in infected versus non-infected tissues using PET/CT scans. | 3 year
  Compare the uptake of [18F]F-TMP in infected versus non-infected tissues using interpretation of PET scan images (using maxSUV and meanSUV of each ROI which will be drawn manually in tissues of interest including but not limited to: Blood pool, heart muscle, brain, thyroid, lymph nodes, lung, liver, kidney, small bowel, large bowel, adrenal gland, pancreas, gall bladder, bone, muscle, and gonads)
Describe the change in biodistribution of uptake of [18F]F-TMP in human patients after therapy. | 3 year
  Describe the change in biodistribution of uptake of [18F]F-TMP in human patients after therapy using interpretation of PET scan images (using maxSUV and meanSUV of each ROI which will be drawn manually in tissues of interest including but not limited to: Blood pool, heart muscle, brain, thyroid, lymph nodes, lung, liver, kidney, small bowel, large bowel, adrenal gland, pancreas, gall bladder, bone, muscle, and gonads)
Describe the change in kinetics of uptake of [18F]F-TMP in human patients after therapy. | 3 year
  Describe the change in kinetics of uptake of [18F]F-TMP in human patients after therapy (using maxSUV and meanSUV of each ROI which will be drawn manually in tissues of interest including but not limited to: Blood pool, heart muscle, brain, thyroid, lymph nodes, lung, liver, kidney, small bowel, large bowel, adrenal gland, pancreas, gall bladder, bone, muscle, and gonads)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pryma, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No